CLINICAL TRIAL: NCT00395148
Title: A Novel Mechanism Mediating Anti-atherosclerotic and Metabolic Actions of HDL Cholesterol
Brief Title: Improving Metabolism With HDL Cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Baker Heart Research Institute (Other)
Responsible Party: Prof Bronwyn Kingwell, Baker IDI Heart & Diabetes Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 175/04
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2006-10

CONDITIONS: Heart Disease; Diabetes
MeSH Terms: conditions — Heart Diseases; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rHDL

SUMMARY:
High levels of good cholesterol (HDL) in our blood decreases our chance of having a heart attack. This relates in part to the role good cholesterol plays in reducing build up of fat in the arteries. However, good cholesterol has many other protective effects. We have recently identified three enzymes (proteins) activated by HDL in cells lining the blood vessels, which may be responsible for some of HDL's protective actions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 65 years
* Free of overt coronary disease
* Body mass index <35 kg.m-2
* Fasting plasma glucose > 7 mmol/L-1
* No major illness

Exclusion Criteria:

* Unable to give informed consent
* Smokers
* Abnormal LFT, U&E, FBE or creatinine

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Metabolic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn A Kingwell, PhD, Principal Investigator — Baker Heart Research Institute
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Result] Hoang A, Drew BG, Low H, Remaley AT, Nestel P, Kingwell BA, Sviridov D. Mechanism of cholesterol efflux in humans after infusion of reconstituted high-density lipoprotein. Eur Heart J. 2012 Mar;33(5):657-65. doi: 10.1093/eurheartj/ehr103. Epub 2011 Apr 15. PMID 21498847
- [Result] Drew BG, Carey AL, Natoli AK, Formosa MF, Vizi D, Reddy-Luthmoodoo M, Weir JM, Barlow CK, van Hall G, Meikle PJ, Duffy SJ, Kingwell BA. Reconstituted high-density lipoprotein infusion modulates fatty acid metabolism in patients with type 2 diabetes mellitus. J Lipid Res. 2011 Mar;52(3):572-81. doi: 10.1194/jlr.P012518. Epub 2011 Jan 11. PMID 21224289
- [Result] Calkin AC, Drew BG, Ono A, Duffy SJ, Gordon MV, Schoenwaelder SM, Sviridov D, Cooper ME, Kingwell BA, Jackson SP. Reconstituted high-density lipoprotein attenuates platelet function in individuals with type 2 diabetes mellitus by promoting cholesterol efflux. Circulation. 2009 Nov 24;120(21):2095-104. doi: 10.1161/CIRCULATIONAHA.109.870709. Epub 2009 Nov 9. PMID 19901191
- [Result] Drew BG, Duffy SJ, Formosa MF, Natoli AK, Henstridge DC, Penfold SA, Thomas WG, Mukhamedova N, de Courten B, Forbes JM, Yap FY, Kaye DM, van Hall G, Febbraio MA, Kemp BE, Sviridov D, Steinberg GR, Kingwell BA. High-density lipoprotein modulates glucose metabolism in patients with type 2 diabetes mellitus. Circulation. 2009 Apr 21;119(15):2103-11. doi: 10.1161/CIRCULATIONAHA.108.843219. Epub 2009 Apr 6. PMID 19349317
- [Result] Patel S, Drew BG, Nakhla S, Duffy SJ, Murphy AJ, Barter PJ, Rye KA, Chin-Dusting J, Hoang A, Sviridov D, Celermajer DS, Kingwell BA. Reconstituted high-density lipoprotein increases plasma high-density lipoprotein anti-inflammatory properties and cholesterol efflux capacity in patients with type 2 diabetes. J Am Coll Cardiol. 2009 Mar 17;53(11):962-71. doi: 10.1016/j.jacc.2008.12.008. PMID 19281927